CLINICAL TRIAL: NCT03384693
Title: A Pilot Trial of Using Pre-Transplant Risk Stratification and Prophylactic Defibrotide to Prevent Serious Thrombotic Microangiopathy in High-Risk Hematopoietic Stem Cell Transplant Patients
Brief Title: Defibrotide TMA Prophylaxis Pilot Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-23356
Record Dates: First submitted 2017-12-11; First posted 2017-12-27 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Thrombotic Microangiopathies
Keywords: hematopoeitic stem cell transplant; prophylactic defibrotide
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — defibrotide

STUDY DESIGN:
Intervention Model Description: Defibrotide 6.25mg/kg administered intravenously for 28-35 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Prophylactic Defibrotide (Experimental): 6.25mg/kg administered intravenously every 6 hours for 28 to 35 days, starting on the day before conditioning is initiated.
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — Defibrotide is an anticoagulant and fibrinolytic agent that has been shown to be an effective treatment in other endothelial disorders such as hepatic veno-occlusive disease.
  Other Names: Defitelio

SUMMARY:
Thrombotic microangiopathy (TMA) is a common complication in the stem cell transplant population. Certain populations within the hematopoietic stem cell transplant (HSCT) population are at a higher risk than others. Defibrotide is an endothelial stabilizing agent which may prevent the endothelial damage that triggers TMA in HSCT patients. The feasibility, safety, and efficacy of defibrotide prophylaxis in a pediatric transplant population is unknown. Twenty five patients age 0 to 30 years receiving autologous or allogeneic hematopoeitic stem cell transplant who meet TMA high risk criteria will be enrolled. Patients will receive Defibrotide for 28-35 days starting before conditioning, and will be closely monitored for any adverse events up through 6 months post-transplant. The feasibility of administering defibrotide will be evaluated as well as incidence of TMA.

DETAILED DESCRIPTION:
This is an open-label, single arm pilot study of defibrotide given as prophylaxis to patients receiving a conditioned stem cell transplant for the purpose of preventing post-transplant microangiopathy. The University of California San Francisco Blood and Marrow Transplant program reviewed all cases of non-relapse related death from 2012 through 2015 and identified a complication of endothelial injury known as transplant associated thrombotic microangiopathy (TMA) as the most common cause of transplant related mortality in its patient population. TMA is a multi-system disease in which widespread endothelial injury leads to microangiopathic hemolytic anemia, intravascular platelet activation and formation of thrombi within the microcirculation. Diagnosis of TMA can be difficult as systemic signs and symptoms of TMA are often similar to other common transplant complications, such as medication induced hypertension and cytopenias. The reported prevalence of TMA is varied likely due to diagnostic uncertainty and transplant center expertise, but large retrospective studies have reported it as 10-39%, with the majority of cases occurring in the first 100 days after transplant. Of the patients who develop TMA, approximately half of them will develop severe disease. Outcomes are poor with a reported 30-50% mortality rate and as high as 80% in patients with severe disease. Furthermore, survivors of TMA may have significant morbidity (e.g. renal failure and need for long-term dialysis, heart failure, and significantly prolonged hospital admission). There is no gold standard of treatment for TMA. Supportive care includes renal support, discontinuation of calcineurin inhibitors, and treatment of infections. Treatment options include plasma exchange, complement cascade blockade, and defibrotide. Early treatment is crucial to decrease morbidity and mortality.

Despite the early recognition and treatment of TMA, poor outcomes occur when patients are treated with complement blockade alone. This suggests that complement activation may trigger a complex cascade of parallel inflammatory mediators that lead to end organ damage independent of the complement pathway. The goal is to prevent TMA whenever possible via augmentation of endothelial repair. Defibrotide is an anticoagulant and fibrinolytic agent that has been shown to be an effective treatment in other endothelial disorders such as hepatic veno-occlusive disease. It is a polydeoxyribonucleotide salt that blocks plasminogen activator inhibitor-1 (PAI-1) and attenuates the effect of tumor necrosis factor. It also increases prostaglandin E2 and prostacyclin levels which alters the platelet activity adhesion and aggregation and relaxes the smooth muscle of blood vessel walls. All of this likely protects the endothelium from damage. It has been shown that patients with TMA who were treated with defibrotide had a 77% response rate.

The use of defibrotide in the context of veno occlusive disease (VOD) treatment and prevention has been studied extensively, including a landmark report showing that defibrotide given to children during stem cell transplant conditioning is safe and effective in the prevention of veno-occlusive disease. Also, defibrotide showed a 67-77% response rate when used as treatment in patients who developed TMA. However, there has not been a prospective study to show that such prophylaxis is effective in the prevention of TMA in pediatric patients undergoing hematopoetic stem cell transplant (HCT).

Patients will receive Defibrotide 6.25mg/kg via two hour intravenous infusions given every 6 hours. Defibrotide will start the day before conditioning is initiated, and will last for 28 to 35 days. During defibrotide administration, participants will have assessments of administration feasibility, hypersensitivity reaction, and bleeding. All hematopoietic stem cell transplant standard of care evaluations will be conducted, including routine clinical evaluations and laboratory assessments.

Patients will be followed for 6 months post-HSCT, or until death, whichever occurs first. All patients will be evaluated for toxicity from the time of their first treatment with the study drug. The study will use the CTCAE v4.03 for reporting of non-hematologic adverse events and modified criteria for hematologic adverse events. Patients removed from study for unacceptable treatment related adverse event(s) will be followed until resolution or stabilization of all treatment-related adverse events to Grade 2 or lower.

Biomarkers indicative of endothelial damage and TMA activity will be drawn to assess subclinical TMA activity as well as risk for subsequent development of TMA while on defibrotide. These include plasma free hemoglobin, suppression of tumorigenicity, angiopoietin 2, and plasminogen activator inhibitor - 1. Study labs will be assessed at 4 time points prior to Day +21, and at diagnosis of TMA.

ELIGIBILITY:
Inclusion Criteria

1. Age 0-30 years of age
2. Life expectancy > 6 months
3. Eastern Cooperative Oncology Group or Karnofsky Performance Status >40
4. Meets minimum organ function requirements per institutional standard of care guiding clearance for autologous or allogeneic stem cell transplantation.
5. Patients must meet TMA High-Risk criteria 5A or 5B below:

5A. Patients undergoing tandem autologous transplant with thiotepa in one or more of the conditioning regimens

OR:

5B. . Patients with at least 3 of the following characteristics:

1. >10 years of age
2. Non-Caucasian race/ Hispanic ethnicity
3. Undergoing haploidentical transplant
4. Minor ABO blood group mismatch

Exclusion Criteria:

1. Age >30 years
2. Life expectancy < 6 months
3. Known bleeding diathesis or bleeding risk deemed by the treating physician to be a contraindication to administration of anticoagulants.
4. Known hypersensitivity reaction to defibrotide
5. Any patient not meeting TMA High-Risk criteria
6. Pregnant women are excluded from this study because they will be receiving teratogenic therapy as part of the stem cell transplant.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Higham, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Benioff Children's Hospital at UCSF Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in scientific journals after de-identification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers can submit a request for access to the study Steering Committee. If the proposal is determined to be methodologically sound, data requestors will need to sign a data access agreement prior to gaining access.

REFERENCES:
- [Background] Cho BS, Yahng SA, Lee SE, Eom KS, Kim YJ, Kim HJ, Lee S, Min CK, Cho SG, Kim DW, Lee JW, Min WS, Park CW. Validation of recently proposed consensus criteria for thrombotic microangiopathy after allogeneic hematopoietic stem-cell transplantation. Transplantation. 2010 Oct 27;90(8):918-26. doi: 10.1097/TP.0b013e3181f24e8d. PMID 20717073
- [Background] Choi CM, Schmaier AH, Snell MR, Lazarus HM. Thrombotic microangiopathy in haematopoietic stem cell transplantation: diagnosis and treatment. Drugs. 2009;69(2):183-98. doi: 10.2165/00003495-200969020-00004. PMID 19228075
- [Background] Corbacioglu S, Cesaro S, Faraci M, Valteau-Couanet D, Gruhn B, Rovelli A, Boelens JJ, Hewitt A, Schrum J, Schulz AS, Muller I, Stein J, Wynn R, Greil J, Sykora KW, Matthes-Martin S, Fuhrer M, O'Meara A, Toporski J, Sedlacek P, Schlegel PG, Ehlert K, Fasth A, Winiarski J, Arvidson J, Mauz-Korholz C, Ozsahin H, Schrauder A, Bader P, Massaro J, D'Agostino R, Hoyle M, Iacobelli M, Debatin KM, Peters C, Dini G. Defibrotide for prophylaxis of hepatic veno-occlusive disease in paediatric haemopoietic stem-cell transplantation: an open-label, phase 3, randomised controlled trial. Lancet. 2012 Apr 7;379(9823):1301-9. doi: 10.1016/S0140-6736(11)61938-7. Epub 2012 Feb 23. PMID 22364685
- [Background] Corti P, Uderzo C, Tagliabue A, Della Volpe A, Annaloro C, Tagliaferri E, Balduzzi A. Defibrotide as a promising treatment for thrombotic thrombocytopenic purpura in patients undergoing bone marrow transplantation. Bone Marrow Transplant. 2002 Mar;29(6):542-3. doi: 10.1038/sj.bmt.1703414. No abstract available. PMID 11960280
- [Background] Jodele S, Dandoy CE, Myers KC, El-Bietar J, Nelson A, Wallace G, Laskin BL. New approaches in the diagnosis, pathophysiology, and treatment of pediatric hematopoietic stem cell transplantation-associated thrombotic microangiopathy. Transfus Apher Sci. 2016 Apr;54(2):181-90. doi: 10.1016/j.transci.2016.04.007. Epub 2016 Apr 25. PMID 27156964
- [Background] Jodele S, Davies SM, Lane A, Khoury J, Dandoy C, Goebel J, Myers K, Grimley M, Bleesing J, El-Bietar J, Wallace G, Chima RS, Paff Z, Laskin BL. Diagnostic and risk criteria for HSCT-associated thrombotic microangiopathy: a study in children and young adults. Blood. 2014 Jul 24;124(4):645-53. doi: 10.1182/blood-2014-03-564997. Epub 2014 May 29. PMID 24876561
- [Background] Jodele S, Zhang K, Zou F, Laskin B, Dandoy CE, Myers KC, Lane A, Meller J, Medvedovic M, Chen J, Davies SM. The genetic fingerprint of susceptibility for transplant-associated thrombotic microangiopathy. Blood. 2016 Feb 25;127(8):989-96. doi: 10.1182/blood-2015-08-663435. Epub 2015 Nov 24. PMID 26603840
- [Background] Kim SS, Patel M, Yum K, Keyzner A. Hematopoietic stem cell transplant-associated thrombotic microangiopathy: review of pharmacologic treatment options. Transfusion. 2015 Feb;55(2):452-8. doi: 10.1111/trf.12859. Epub 2014 Sep 11. PMID 25209960
- [Background] Kojouri K, George JN. Thrombotic microangiopathy following allogeneic hematopoietic stem cell transplantation. Curr Opin Oncol. 2007 Mar;19(2):148-54. doi: 10.1097/CCO.0b013e3280148a2f. PMID 17272988
- [Background] Laskin BL, Goebel J, Davies SM, Jodele S. Small vessels, big trouble in the kidneys and beyond: hematopoietic stem cell transplantation-associated thrombotic microangiopathy. Blood. 2011 Aug 11;118(6):1452-62. doi: 10.1182/blood-2011-02-321315. Epub 2011 May 19. PMID 21596850
- [Background] Obut F, Kasinath V, Abdi R. Post-bone marrow transplant thrombotic microangiopathy. Bone Marrow Transplant. 2016 Jul;51(7):891-7. doi: 10.1038/bmt.2016.61. Epub 2016 Mar 14. PMID 26974272
- [Background] Richardson PG, Murakami C, Jin Z, Warren D, Momtaz P, Hoppensteadt D, Elias AD, Antin JH, Soiffer R, Spitzer T, Avigan D, Bearman SI, Martin PL, Kurtzberg J, Vredenburgh J, Chen AR, Arai S, Vogelsang G, McDonald GB, Guinan EC. Multi-institutional use of defibrotide in 88 patients after stem cell transplantation with severe veno-occlusive disease and multisystem organ failure: response without significant toxicity in a high-risk population and factors predictive of outcome. Blood. 2002 Dec 15;100(13):4337-43. doi: 10.1182/blood-2002-04-1216. Epub 2002 Aug 1. PMID 12393437
- [Background] Rosenthal J. Hematopoietic cell transplantation-associated thrombotic microangiopathy: a review of pathophysiology, diagnosis, and treatment. J Blood Med. 2016 Sep 2;7:181-6. doi: 10.2147/JBM.S102235. eCollection 2016. PMID 27621680
- [Background] Uderzo C, Bonanomi S, Busca A, Renoldi M, Ferrari P, Iacobelli M, Morreale G, Lanino E, Annaloro C, Volpe AD, Alessandrino P, Longoni D, Locatelli F, Sangalli H, Rovelli A. Risk factors and severe outcome in thrombotic microangiopathy after allogeneic hematopoietic stem cell transplantation. Transplantation. 2006 Sep 15;82(5):638-44. doi: 10.1097/01.tp.0000230373.82376.46. PMID 16969286
- [Background] Uderzo C, Fumagalli M, De Lorenzo P, Busca A, Vassallo E, Bonanomi S, Lanino E, Dini G, Varotto S, Messina C, Miniero R, Valsecchi MG, Balduzzi A. Impact of thrombotic thrombocytopenic purpura on leukemic children undergoing bone marrow transplantation. Bone Marrow Transplant. 2000 Nov;26(9):1005-9. doi: 10.1038/sj.bmt.1702648. PMID 11100281
- [Background] Wingard JR, Majhail NS, Brazauskas R, Wang Z, Sobocinski KA, Jacobsohn D, Sorror ML, Horowitz MM, Bolwell B, Rizzo JD, Socie G. Long-term survival and late deaths after allogeneic hematopoietic cell transplantation. J Clin Oncol. 2011 Jun 1;29(16):2230-9. doi: 10.1200/JCO.2010.33.7212. Epub 2011 Apr 4. PMID 21464398
- [Background] Yeates L, Slatter MA, Bonanomi S, Lim FLWI, Ong SY, Dalissier A, Barberi W, Shulz A, Duval M, Heilmann C, Willekens A, Hwang WHY, Uderzo C, Bader P, Gennery AR. Use of defibrotide to treat transplant-associated thrombotic microangiopathy: a retrospective study of the Paediatric Diseases and Inborn Errors Working Parties of the European Society of Blood and Marrow Transplantation. Bone Marrow Transplant. 2017 May;52(5):762-764. doi: 10.1038/bmt.2016.351. Epub 2017 Jan 16. No abstract available. PMID 28092354
- [Derived] Higham CS, Shimano KA, Melton A, Kharbanda S, Chu J, Dara J, Winestone LE, Hermiston ML, Huang JN, Dvorak CC. A pilot trial of prophylactic defibrotide to prevent serious thrombotic microangiopathy in high-risk pediatric patients. Pediatr Blood Cancer. 2022 May;69(5):e29641. doi: 10.1002/pbc.29641. Epub 2022 Mar 6. PMID 35253361

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prophylactic Defibrotide
Started | 25
Completed | 22
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: 25 patients who started therapy
Arm/Group | Prophylactic Defibrotide
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 2
  Unknown or Not Reported | 0
Diagnosis [Count of Participants; unit: Participants]
  Leukemia | 9
  Lymphoma | 2
  Neuroblastoma | 14
Recipient CMV (cytomegalovirus) serostatus [Count of Participants; unit: Participants]
  Positive | 14
  Negative | 11
Donor type [Count of Participants; unit: Participants]
  Unrelated | 1
  Haploidentical | 10
  N/A (Autologous) | 14
MIBG (Metaiodobenzylguanidine) therapy prior to transplant [Count of Participants; unit: Participants]
  Yes | 4
  No | 21
Conditioning backbone [Count of Participants; unit: Participants]
  TBI based | 3
  Melphalan based | 6
  Busulfan based | 2
  Other (Autologous) | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent of Total Doses of Defibrotide That Were Missed [Feasibility]
Description: Feasibility will be determined with regard to administration concurrently with chemotherapy and supportive medications before, during, and after stem cell infusion.
Time Frame: From first treatment with study drug to day +21 post Transplant
Measure: Median (Full Range); unit: percentage of missed doses
Arm/Group | Prophylactic Defibrotide
Number analyzed (Participants) | 22
percentage of missed doses | 0.7 [0.5 to 2.0]

2. Primary Outcome: Participants With Reportable Serious Adverse Events [Safety] Per CTACAE v5 Grade 3 or Higher
Description: Safety was assessed by evaluating drug-related Serious Adverse Events per CTACAE v5 that occur after prophylactic administration of defibrotide. Analyses will be performed for all patients having received at least one dose of study drug.
Time Frame: From first treatment with study drug to 6 months post-transplant
Population: all patients having received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Defibrotide
Number analyzed (Participants) | 25
Participants | 3

3. Primary Outcome: Participants With Clinically Significant Bleeding Requiring Discontinuation of Therapy [Safety]
Description: Bleeding was assessed using Common Toxicity Criteria for Adverse Events version 4.03. (CTCAE). Study drug was permanently discontinued at grade 3 bleeding or higher. Analyses will be performed for all patients having received at least one dose of study drug.
Time Frame: From first treatment with study drug to 6 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Defibrotide
Number analyzed (Participants) | 25
Participants | 3

4. Primary Outcome: Participants With Hypersensitivity Reaction Requiring Discontinuation of Therapy [Safety]
Description: Hypersensitivity reaction will be assessed using Common Toxicity Criteria for Adverse Events version 4.03.
  For grade 2 hypersensitivity reaction, study drug will be held until it resolves to grade 1 or lower. Study drug will be permanently discontinued at grade 3 hypersensitivity reaction or higher. Analyses will be performed for all patients having received at least one dose of study drug.
Time Frame: From first treatment with study drug to 6 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Defibrotide
Number analyzed (Participants) | 25
Participants | 3

5. Secondary Outcome: Number of Patients With TMA Enrolled on the Study
Description: Evidence of microangiopathy, with either clinical markers/organ dysfunction or presence of biomarkers, or one of the following: 1) presence of schistocytes in peripheral blood; 2) Histologic evidence of microangiopathy on a tissue specimen; 3) Undetectable haptoglobin with increased reticulocyte counts. If there is no evidence of microangiopathy but at least one clinical marker or at least 3 biomarkers, the participant will meet the criteria for TMA incidence.
  Based on prior analysis at our center, we anticipated an incidence of TA-TMA of 28.2% (95 CI, 17.8-38.6%) in the high-risk patients undergoing allogeneic transplants and 40% (95% CI, 13.9-69.5%) in the neuroblastoma patients undergoing planned tandem HSCT
Time Frame: 6 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Defibrotide
Number analyzed (Participants) | 25
Participants | 1

6. Secondary Outcome: Number of Patients With Severe TMA
Description: Severe TMA is defined as any TMA meeting the criteria in Objective 2 with the following complications: renal dysfunction requiring dialysis, pleural or pericardial effusion requiring any medical or surgical intervention, central nervous system dysfunction including seizure or posterior reversible encephalopathy syndrome, or death.
Time Frame: 6 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Defibrotide
Number analyzed (Participants) | 25
Participants | 0

7. Other Pre Specified Outcome: Incidence of Elevation of Single or Combination of Biomarkers Predictive of Development of TMA
Description: Values will be analyzed to determine whether any one biomarker or a combination of biomarkers may be predictive of TMA development or severity.
Time Frame: 6 months post-transplant
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Incidence of TMA
Description: Evidence of microangiopathy, with either clinical markers/organ dysfunction or presence of biomarkers, or one of the following: 1) presence of schistocytes in peripheral blood; 2) Histologic evidence of microangiopathy on a tissue specimen; 3) Undetectable haptoglobin with increased reticulocyte counts. If there is no evidence of microangiopathy but at least one clinical marker or at least 3 biomarkers, the participant will meet the criteria for TMA incidence.
Time Frame: Day 30, day 100 and day 180 post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Defibrotide
Number analyzed (Participants) | 25
Participants
  Day 30 | 1
  day 100 | 0
  Day 180 | 0

9. Other Pre Specified Outcome: Non Relapse Mortality
Description: Deaths which cannot be attributed to disease relapse or progression
Time Frame: Day 100 and day 180 post-transplant
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Prophylactic Defibrotide
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylactic Defibrotide (N=25)
Bleeding (General disorders) | 3

LIMITATIONS AND CAVEATS:
Limitations include:

Small single institution non-randomized trial. Combination of two separate patient populations at high-risk for TA-TMA allowed for a more robust study, but smaller numbers of patients in each of the groups limits sub-analysis.

Some interesting preliminary findings with study biomarkers but the study is too small to draw definitive conclusions regarding utility.

No current CLIA-approved lab measuring ANG-2, limiting applicability of this test to the clinical setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT03384693/Prot_SAP_000.pdf